CLINICAL TRIAL: NCT05124678
Title: A Phase II Trial to Describe the Pharmacokinetics, Safety and Efficacy of Pharmacogenetics-guided Dosing of Isoniazid in Patients With HIV-associated TB
Brief Title: Pharmacogenetics-guided Isoniazid Dosing in TB-HIV
Acronym: PHINX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDI SRC Ref:16/2020
Record Dates: First submitted 2021-10-01; First posted 2021-11-18 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-10

CONDITIONS: Tuberculosis
Keywords: Pharmacokinetics; Pharmacogenetics; High-dose Isoniazid
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast/intermediate acetylators (Experimental): Participants in this arm have fast/intermediate acetylator status from NAT2 genotyping.
  In the Intensive phase (Month 1-2) of treatment, they will receive; Oral Isoniazid 10mg/kg/day + Rifampicin, Ethambutol and Pyrazinamide at standard dose.
  In the continuation phase (Month 3 - 6 ) of treatment, they will receive; Oral Isoniazid 5mg/kg/day +Rifampicin at standard dose
  Interventions: Drug: Isoniazid Tablets
- Slow acetylators (No Intervention): Participants in this arm have a slow acetylator status from NAT2 genotyping. They will receive the standard of care. In the Intensive phase (Month 1-2) of treatment, they will receive; Oral Isoniazid 5mg/kg/day + Rifampicin, Ethambutol and Pyrazinamide at standard dose.
  In the continuation phase (Month 3 - 6 ) of treatment, they will receive; Oral Isoniazid 5mg/kg/day +Rifampicin at standard dose

INTERVENTIONS:
Drug: Isoniazid Tablets — High dose of isoniazid
  Other Names: INH
  Arms: Fast/intermediate acetylators

SUMMARY:
The current TB treatment as recommended by World Health Organization (WHO) although capable of achieving 85% cure rates, has limitations, in particular drug interactions, toxicities, and the long treatment duration which increases the possibility of nonadherence.

Sub-therapeutic isoniazid concentrations were demonstrated in several studies, including our previous work, carried out among patients with tuberculosis receiving the standard dose (5mg/kg) of isoniazid. The investigators found 78% of patients with HIV had isoniazid concentrations below the recommended threshold. Malabsorption, drug-drug interactions, poor adherence due to high pill burden may contribute to this. Pharmacogenetic variation may compound these factors; isoniazid displays inter-individual variation in serum concentrations and clearance due to differences in individual acetylator status.

While patients who metabolize isoniazid slowly (slow acetylators) are at a higher risk of high drug concentrations and toxicities, fast acetylators are more likely to have sub-therapeutic isoniazid concentrations.

In other studies, insufficient exposure with isoniazid, one of the cornerstone drugs for TB treatment, has been associated with delayed sputum clearance, development of drug resistance, and treatment failure.

Isoniazid is metabolized by the enzyme N-acetyl transferase, which in turn is controlled by the N-acetyl transferase-2 (NAT-2) gene. Polymorphisms in this gene are responsible for the N-acetylation phenotypes, with the distribution of NAT-2 fast, intermediate, and slow acetylators being highly variable especially among African populations.

Given that NAT2 acetylator status explains most of the variability in INH exposures, knowledge of NAT2 status may be a simpler way to select the right dose for individual patients. The investigators will therefore provide higher doses to fast acetylators and compare the isoniazid pharmacokinetics in these patients to slow acetylators who receive the standard dose, who are more likely to already be achieving target concentrations.

DETAILED DESCRIPTION:
N-acetyl transferase genotyping will be performed on HIV infected patients diagnosed with T B. Slow acetylators will be initiated on the standard dose of isoniazid (5mg/kg) while fast and intermediate acetylators will be initiated on 10mg/kg of isoniazid. All other TB drugs will be given at their standard doses.

Monitoring for toxicities will be performed every two weeks (including ALT and screening for peripheral neuropathy) and isoniazid concentrations will be measured four weeks after initiating treatment at Ohr, 30mins, 1 hr, Thr and 4hr following observed drug intake.

Patients will be continued on standard dose isoniazid after completing the first 8 weeks of treatment (intensive phase).

Sputum cultures for mycobacteria will be performed at baseline, week 2, 4 and week 8. TB treatment outcome will be assessed after 6 months of treatment.

Non-linear mixed effects modelling will be used to model PK-PD data taking into account clinical and demographic factors like age, sex and BMI. The investigators will develop a model to establish the population parameters for isoniazid (for example clearance, absorption rate constant and volume of distribution) and the variability around these primary PK parameters. The investigators will then use the model to derive secondary PK parameters, namely area under the concentration-time curve (AUC) and maximum concentrations (Cmax) of isoniazid for each participant. The investigators will compare the PK parameters of isoniazid in fast/intermediate acetylators taking 10mg/kg and slow acetylators taking 5mg/kg of isoniazid.

In addition to the main objectives of the study, the investigators will also compare the PK in patients in the PG guided isoniazid dosing group to those in the historical cohort while matching for NAT2 status, age and sex. In the historical cohort, NAT-2 acetlyator genotyping was performed but patients received standard dosing regardless of NAT-2 acetylator status. In this trial, the investigators will use pharmacogenetic guided therapy for all participants. The investigators will therefore be able to compare the pharmacokinetic data above, safety and efficacy in patients who received pharmacogenetic therapy and those who did not.

The investigators will use PK-PD models to describe the relationship between concentrations and pharmacodynamic data (including toxicities and sputum conversion at week 8) in patients on the different doses. In addition to this, the investigators will also make this same comparison for patients in this study and those who did not receive PG guided therapy from the historical cohort. The investigators will also compare the number of grade 3-5 adverse events and time to sputum culture conversion in patients in patients who did and did not receive PG guided therapy while matching for NAT2 status, age and sex

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Age of ≥18 years
* Bacteriologically confirmed pulmonary TB (determined by Xpert, culture, or microscopy)
* Confirmed HIV-1 infection.
* On TB treatment for ≤ 7 days at the time of enrolment (Within this time, the patient is still expected to have mycobacteria present in sputum and will provide enough time to conduct screening procedures)

Exclusion Criteria:

* TB infection of any organ/systems requiring TB treatment longer than 6 months
* Pregnancy
* Decompensated liver disease and/or aminotransferases >2.5 x ULN

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Estimate the maximum concentrations of isoniazid stratified by NAT2 group | Week 4 of treatment
  Maximum concentrations (Cmax)
Estimate the area under the concentration-time curve of isoniazid stratified by NAT2 group | Week 4 of treatment
  Area under the concentration-time curve (AUC)
Estimate the of Clearance isoniazid stratified by NAT2 group | Week 4 of treatment
  Clearance (L/h)
Estimate the Volume of distribution of isoniazid stratified by NAT2 group | Week 4 of treatment
  Volume of distribution (L)

SECONDARY OUTCOMES:
Drug-induced hepatotoxicity | Up to week 8 of treatment
  Grade 2 or higher elevation in ALT or total bilirubin (drug-induced hepatotoxicity)
Other drug-related adverse events | Up to week 8 of treatment
  Other grade 2 or higher adverse events
Peripheral neuropathy | Up to week 8 of treatment
  Grade 2 or higher peripheral neuropathy
Sputum culture conversion at week 8 | Up to week 8 of treatment
  Proportion of patients who remain sputum positive

CONTACTS AND LOCATIONS:
Overall Officials: Christine Sekaggya-Wiltshire, MBChB, PhD, Principal Investigator — Infectious Diseases Institute-Kampala
Locations (1):
- Infectious Diseases Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data (IPD) will made available to other researchers for further analysis or met-analysis upon reasonable request to the investigators.
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after publication of study results.
Access Criteria: A direct request shall be made to the investigators .

REFERENCES:
- [Background] Adams LV, Mahlalela N, Talbot EA, Pasipamire M, Ginindza S, Calnan M, Haumba S. High completion rates of isoniazid preventive therapy among persons living with HIV in Swaziland. Int J Tuberc Lung Dis. 2017 Oct 1;21(10):1127-1132. doi: 10.5588/ijtld.16.0946. PMID 28911356
- [Background] World Health Organization, Guildelines for treatment of Tuberculosis. 2013.
- [Background] Han T. Effectiveness of standard short-course chemotherapy for treating tuberculosis and the impact of drug resistance on its outcome. JBI Libr Syst Rev. 2006;4(3):1-27. doi: 10.11124/01938924-200604030-00001. PMID 27819814
- [Background] Chideya S, Winston CA, Peloquin CA, Bradford WZ, Hopewell PC, Wells CD, Reingold AL, Kenyon TA, Moeti TL, Tappero JW. Isoniazid, rifampin, ethambutol, and pyrazinamide pharmacokinetics and treatment outcomes among a predominantly HIV-infected cohort of adults with tuberculosis from Botswana. Clin Infect Dis. 2009 Jun 15;48(12):1685-94. doi: 10.1086/599040. PMID 19432554
- [Background] McIlleron H, Rustomjee R, Vahedi M, Mthiyane T, Denti P, Connolly C, Rida W, Pym A, Smith PJ, Onyebujoh PC. Reduced antituberculosis drug concentrations in HIV-infected patients who are men or have low weight: implications for international dosing guidelines. Antimicrob Agents Chemother. 2012 Jun;56(6):3232-8. doi: 10.1128/AAC.05526-11. Epub 2012 Mar 12. PMID 22411614
- [Background] Park JS, Lee JY, Lee YJ, Kim SJ, Cho YJ, Yoon HI, Lee CT, Song J, Lee JH. Serum Levels of Antituberculosis Drugs and Their Effect on Tuberculosis Treatment Outcome. Antimicrob Agents Chemother. 2015 Oct 12;60(1):92-8. doi: 10.1128/AAC.00693-15. Print 2016 Jan. PMID 26459901
- [Background] Peloquin CA, Nitta AT, Burman WJ, Brudney KF, Miranda-Massari JR, McGuinness ME, Berning SE, Gerena GT. Low antituberculosis drug concentrations in patients with AIDS. Ann Pharmacother. 1996 Sep;30(9):919-25. doi: 10.1177/106002809603000901. PMID 8876848
- [Background] Sekaggya-Wiltshire C, von Braun A, Lamorde M, Ledergerber B, Buzibye A, Henning L, Musaazi J, Gutteck U, Denti P, de Kock M, Jetter A, Byakika-Kibwika P, Eberhard N, Matovu J, Joloba M, Muller D, Manabe YC, Kamya MR, Corti N, Kambugu A, Castelnuovo B, Fehr JS. Delayed Sputum Culture Conversion in Tuberculosis-Human Immunodeficiency Virus-Coinfected Patients With Low Isoniazid and Rifampicin Concentrations. Clin Infect Dis. 2018 Aug 16;67(5):708-716. doi: 10.1093/cid/ciy179. PMID 29514175
- [Background] Ding J, Thuy Thuong Thuong N, Pham TV, Heemskerk D, Pouplin T, Tran CTH, Nguyen MTH, Nguyen PH, Phan LP, Nguyen CVV, Thwaites G, Tarning J. Pharmacokinetics and Pharmacodynamics of Intensive Antituberculosis Treatment of Tuberculous Meningitis. Clin Pharmacol Ther. 2020 Apr;107(4):1023-1033. doi: 10.1002/cpt.1783. Epub 2020 Feb 29. PMID 31956998
- [Background] Jindani A, Aber VR, Edwards EA, Mitchison DA. The early bactericidal activity of drugs in patients with pulmonary tuberculosis. Am Rev Respir Dis. 1980 Jun;121(6):939-49. doi: 10.1164/arrd.1980.121.6.939. No abstract available. PMID 6774638
- [Background] Sloan D: Pharmacokinetic Variability in TB Therapy: Associations with HIV and Effect on Outcome. In: Conference on Retroviruses and Opportunistic Infections. Boston, Massachusetts, U.S.A; 2014
- [Background] Mah A, Kharrat H, Ahmed R, Gao Z, Der E, Hansen E, Long R, Kunimoto D, Cooper R. Serum drug concentrations of INH and RMP predict 2-month sputum culture results in tuberculosis patients. Int J Tuberc Lung Dis. 2015 Feb;19(2):210-5. doi: 10.5588/ijtld.14.0405. PMID 25574921
- [Background] Cordes H, Thiel C, Aschmann HE, Baier V, Blank LM, Kuepfer L. A Physiologically Based Pharmacokinetic Model of Isoniazid and Its Application in Individualizing Tuberculosis Chemotherapy. Antimicrob Agents Chemother. 2016 Sep 23;60(10):6134-45. doi: 10.1128/AAC.00508-16. Print 2016 Oct. PMID 27480867
- [Background] Katiyar SK, Bihari S, Prakash S, Mamtani M, Kulkarni H. A randomised controlled trial of high-dose isoniazid adjuvant therapy for multidrug-resistant tuberculosis. Int J Tuberc Lung Dis. 2008 Feb;12(2):139-45. PMID 18230245
- [Background] Sekaggya-Wiltshire C, von Braun A, Scherrer AU, Manabe YC, Buzibye A, Muller D, Ledergerber B, Gutteck U, Corti N, Kambugu A, Byakika-Kibwika P, Lamorde M, Castelnuovo B, Fehr J, Kamya MR. Anti-TB drug concentrations and drug-associated toxicities among TB/HIV-coinfected patients. J Antimicrob Chemother. 2017 Apr 1;72(4):1172-1177. doi: 10.1093/jac/dkw534. PMID 28108678
- [Background] Denti P, Jeremiah K, Chigutsa E, Faurholt-Jepsen D, PrayGod G, Range N, Castel S, Wiesner L, Hagen CM, Christiansen M, Changalucha J, McIlleron H, Friis H, Andersen AB. Pharmacokinetics of Isoniazid, Pyrazinamide, and Ethambutol in Newly Diagnosed Pulmonary TB Patients in Tanzania. PLoS One. 2015 Oct 26;10(10):e0141002. doi: 10.1371/journal.pone.0141002. eCollection 2015. PMID 26501782
- [Background] Aklillu E, Carrillo JA, Makonnen E, Bertilsson L, Djordjevic N. N-Acetyltransferase-2 (NAT2) phenotype is influenced by genotype-environment interaction in Ethiopians. Eur J Clin Pharmacol. 2018 Jul;74(7):903-911. doi: 10.1007/s00228-018-2448-y. Epub 2018 Mar 27. PMID 29589062
- [Background] Zaid RB, Nargis M, Neelotpol S, Sayeed MA, Banu A, Shurovi S, Hassan KN, Salimullah M, Ali L, Azad Khan AK. Importance of acetylator phenotype in the identity of Asian populations. Hum Biol. 2007 Jun;79(3):363-8. doi: 10.1353/hub.2007.0041. PMID 18078208
- [Background] Meier C, Brauchli YB, Jick SS, Kraenzlin ME, Meier CR. Use of depot medroxyprogesterone acetate and fracture risk. J Clin Endocrinol Metab. 2010 Nov;95(11):4909-16. doi: 10.1210/jc.2010-0032. Epub 2010 Aug 4. PMID 20685865
- [Background] Burhan E, Ruesen C, Ruslami R, Ginanjar A, Mangunnegoro H, Ascobat P, Donders R, van Crevel R, Aarnoutse R. Isoniazid, rifampin, and pyrazinamide plasma concentrations in relation to treatment response in Indonesian pulmonary tuberculosis patients. Antimicrob Agents Chemother. 2013 Aug;57(8):3614-9. doi: 10.1128/AAC.02468-12. Epub 2013 May 20. PMID 23689725
- [Background] Migliori GB, Raviglione MC, Schaberg T, Davies PD, Zellweger JP, Grzemska M, Mihaescu T, Clancy L, Casali L. Tuberculosis management in Europe. Task Force of the European Respiratory Society (ERS), the World Health Organisation (WHO) and the International Union against Tuberculosis and Lung Disease (IUATLD) Europe Region. Eur Respir J. 1999 Oct;14(4):978-92. doi: 10.1183/09031936.99.14497899. No abstract available. PMID 10573254